CLINICAL TRIAL: NCT05873790
Title: A Prospective Observational Study of MRD Dynamic Monitoring in First-Line Serplulimab Plus Chemotherapy in Treatment of Extensive Small Cell Lung Cancer
Brief Title: Minimal Residual Disease Dynamic Monitoring in First-Line Serplulimab Plus Chemotherapy in Treatment of Extensive Small Cell Lung Cancer: An Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 23K048-001
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: Small Cell Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serplulimab and chemotherapy: Participants receive 6 cycles of first-line Serplulimab plus chemotherapy, And MRD testing was performed before treatment, after 2 cycles of treatment, after 6 cycles of treatment, 6 months after the end of chemotherapy, and 1 year after the end of chemotherapy.
  Interventions: Drug: Serplulimab plus chemotherapy

INTERVENTIONS:
Drug: Serplulimab plus chemotherapy — Serplulimab: 4.5 mg/kg via intravenous infusion on Day 1 of each 21-day cycle. Chemotherapy drugs: etoposide + carboplatin/cisplatin Etoposide: 300 mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for a maximum of 6 cycles.
  Carboplatin: 300 mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for a maximum of 6 cycles.
  Cisplatin: 75 mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for a maximum of 6 cycles.

SUMMARY:
Small cell lung cancer (SCLC) is one of the most aggressive lung cancer subtypes, accounting for approximately 15-20% of total lung cancer cases. Although SCLC is relatively sensitive to chemotherapy, it is highly susceptible to recurrence. The advent of immunotherapy has revolutionized the clinical practice of oncology, and the newly released results of the ASTRUM-005 study have led to the incorporation of Serplulimab into the first-line treatment of extensive-stage SCLC. Although immunotherapy in combination with chemotherapy is currently the most promising regimen, due to the limited understanding of genetic alterations and the marked genetic heterogeneity of SCLC, treatment responsiveness varies greatly. Thus, there is an urgent need to find molecular biomarkers that can effectively predict prognosis and further suggest the effectiveness of this new treatment mode.

Minimal residual disease (MRD) refers to the presence of tumor cells disseminated from the primary lesion to distant organs in patients who lack any clinical or radiological signs of metastasis or residual tumor cells left behind after local therapy that eventually lead to local recurrence. These years, the development of real-time, high-sensitivity liquid biopsy assays have enabled the identification of MRD in individual patients with cancer. Multiple studies have demonstrated that detection of MRD dynamics following definitive therapy for solid cancers is strongly prognostic and has extremely high positive predictive value for risk of recurrence and treatment efficacy.

The aim of this study was to explore the predictive value of MRD dynamics on disease prognosis before and after the first-line treatment of Serplulimab in combination with chemotherapy for extensive-stage SCLC.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 2.
* Have previously untreated and confirmed by histological and imaging examinations as extensive small cell lung cancer
* Adequate organ function and expected survival time ≥ 12 weeks;
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.

Key Exclusion Criteria:

* Presence of mixed carcinoma component on histology.
* Patients with other active malignancies within 5 years prior to enrollment.
* Known active autoimmune diseases.
* Currently participate in an interventional clinical study treatment or have been treated with another drug or investigational device within 4 weeks prior to the first dose.
* Use of immunosuppressive agents within 14 days prior to the first dose of study treatment.
* Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient initially diagnosed with extensive small cell lung cancer at the First Hospital of Jilin University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | One year after the end of chemotherapy
  Defined as the time from the first dose of study drug to tumor progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | One year after the end of chemotherapy
  Defined as the time from the first dose of study drug to death due to any cause.
Objective Response Rate (ORR) | One year after the end of chemotherapy
  Defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Disease-Control Rate (DCR) | One year after the end of chemotherapy
  Defined as the proportion of patients with complete response, partial response, and stable disease.

IPD SHARING:
Plan to Share IPD: No